CLINICAL TRIAL: NCT06305832
Title: Salvage Radiotherapy Combined With Androgen Deprivation Therapy (ADT) With or Without Rezvilutamide in the Treatment of Biochemical Recurrence After Radical Prostatectomy for Prostate Cancer: a Prospective, Multicenter, Randomized Controlled Clinical Study
Brief Title: Salvage Radiotherapy Combined With Androgen Deprivation Therapy (ADT) With or Without Rezvilutamide in the Treatment of Biochemical Recurrence After Radical Prostatectomy for Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, PhD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-120
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; Biochemical Recurrence
Keywords: Prostate cancer; Biochemical recurrence; Rezvilutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezvilutamide +ADT+ SRT (Experimental): Rezvilutamide along with ADT for 6 cycles (28 days for each cycle) in combination with salvage radiation therapy (SRT) according to standard of care
  Interventions: Drug: Rezvilutamide; Drug: Androgen deprivation therapy (ADT); Radiation: SRT
- ADT+ SRT (Other): ADT for 6 cycles (28 days for each cycle) in combination with salvage radiation therapy (SRT) according to standard of care
  Interventions: Drug: Androgen deprivation therapy (ADT); Radiation: SRT

INTERVENTIONS:
Drug: Rezvilutamide — Specifications of 80 mg; orally, once a day
  Other Names: SHR3680
  Arms: Rezvilutamide +ADT+ SRT
Drug: Androgen deprivation therapy (ADT) — Androgen deprivation therapy (ADT), the ADT used by each subject will be determined by the investigator,and the dose and frequency of administration will be consistent with the prescription information
Radiation: SRT — SRT according to standard of care (66.6-72 grays will be delivered to the bed of prostate ,~50.4 grays to the pelvis if needed)

SUMMARY:
To evaluate the efficacy and safety of rezvilutamide in combination with androgen deprivation therapy(ADT) and standard salvage radiation therapy(SRT) or SRT combination with ADT in prostate cancer patients with biochemical recurrence of prostate-specific antigen(PSA) persistence after radical prostatectomy(RP).

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥40 years old, male;
* 2. Postoperative pathology showed prostate adenocarcinoma;
* 3. Postoperative pathological stage pN0 or pNx;
* 4. PSA decline < 0.1ng/ml within 8 weeks after radical prostate cancer surgery for at least 6 months
* 5. Biochemical recurrence (PSA rose twice in a row, with an interval of ≥2 weeks and absolute value > 0.2ng/ml), and traditional imaging (bone scan and CT/MRI scan) did not show local recurrence and distant metastasis.
* 6. Have one or more of the following risk factors:

  * Postoperative CAPRA-S score ≥6 points;
  * The pathological score of radical surgery for prostate cancer was Gleason 8-10;
  * The highest postoperative biochemical recurrence PSA > 0.5ng/ml;
  * Postoperative pathological stage PT3/T4;
  * PSADT < 10 months;
* 7. ECOG status is 0-1;
* 8. Life expectancy greater than 10 years;
* 9. Adequate hematological and organ function tests within 4 weeks prior to the first study treatment, as defined below:

  * Neutrophil count (ANC)≥1.5×10^9/L (no granulocyte colony-stimulating factor for 2 weeks prior to cycle 1, day 1);
  * Platelet count (PLT)≥100×10^9/L (no transfusion within 2 weeks prior to day 1 of cycle 1);
  * Hemoglobin (Hb) ≥90g/L
  * Serum creatinine (Cr)≤1.5×ULN or creatinine clearance > 50ml/min;
  * Total bilirubin (BIL)≤1.5×ULN;
  * Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) level ≤2.5×ULN;
  * International Standardized ratio (INR) ≤1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN;
  * Left ventricular ejection fraction (LVEF) ≥50%;
* 10. The subject is willing and understands to sign the informed consent and is able to comply with the agreement.

Exclusion Criteria:

* 1. Previously received endocrine therapy for prostate cancer (including but not limited to goserrelin, levoprorelin, digarek, bicalutamide, abiraterone acetate, darotamine, apatamide, enzalutamide, etc.) or pelvic radiotherapy;
* 2. Postoperative biochemical recurrence, but PSA more than 2 ng/ml;
* 3. Postoperative pathology contains non-adenocarcinoma components, such as neuroendocrine differentiation or small cell features;
* 4. Is currently participating in or has participated in an investigational drug study;
* 5. Known or suspected allergy to reverumide and reverumide excipients;
* 6. Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors that affect drug use and absorption;
* 7. Have a history of epilepsy, or a medical condition that can induce seizures within the 12 months prior to C1D1 (including a history of transient ischemic attacks, cerebral stroke, traumatic brain injury with disturbance of consciousness requiring hospitalization);
* 8. Active heart disease in the 6 months prior to C1D1, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and medically treatable ventricular arrhythmias;
* 9. Have had any other malignancies within the 3 years prior to C1D1 (except for carcinoma in situ that has been in complete remission and malignancies that the investigator determined to be slowly progressing);
* 10. Granulocyte colony-stimulating factor was used for support 2 weeks before C1D1;
* 11. Blood transfusion within 2 weeks before C1D1;
* 12. Active HBV and HCV infected persons (HBV copy number ≥10^4 copies /mL, HCV copy number ≥10^3 copies /mL);
* 13. A history of immunodeficiency (including HIV positive, other acquired, congenital immunodeficiency diseases) or a history of organ transplantation;
* 14. Male subjects whose partner is a fertile woman refuse surgical sterilization or use of effective contraception during the trial period and for 3 months after the last dose of riverutamide.
* 15. The investigator determines subjects who may affect the conduct of clinical studies, who may not be able to comply with the protocol or cooperate with the protocol, and who pose research risks.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
3-year biochemical progression-free survival | 48 months
  biochemical progression is defined as a confirmed prostate specific antigen (PSA) greater than (>) 0.2 nanogram per milliliter (ng/ml) ( the time interval should be over 2 weeks)

SECONDARY OUTCOMES:
progression-free survival (PFS) | 48 months
  Time from entry to biochemical progression or radiologically confirmed progressive disease or death due to any cause
metastasis-free survival (MFS) | 48 months
  Time from entry to radiologically confirmed metastasis disease or death due to any cause.
percentage of undetectable PSA | 48 months
  percentage of undetectable PSA is defined as the proportion of subjects with a PSA level ≤ 0.1 ng/mL after enrollment
ctDNA-positive rate | 48 months
  ctDNA-positive rate was defined as the number of ctDNA subjects detected in the total enrolled population
ctDNA clearance rate | 48 months
  Defined as the number of patients who were ctDNA-positive at enrollment to ctDNA-negative after treatment as a proportion of ctDNA-positive patients enrolled
Adverse Events | 48 months
  According to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No